CLINICAL TRIAL: NCT02268955
Title: Assessment of the Analgesic Efficacy of Intravenous Ibuprofen in Biliary Colic
Brief Title: Analgesic Efficacy of Intravenous Ibuprofen in Biliary Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valleywise Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-067
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-03

CONDITIONS: Biliary Colic
Keywords: Biliary Colic; Abdominal pain; Intravenous Ibuprofen
MeSH Terms: conditions — Abdominal Pain | interventions — Ibuprofen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group: Adults age 18-55 years (Placebo Comparator): Saline-only control group
  Interventions: Drug: Saline
- IV Ibuprofen: Adults age 18-55 years (Active Comparator): Patients receiving intravenous ibuprofen therapy
  Interventions: Drug: IV Ibuprofen

INTERVENTIONS:
Drug: IV Ibuprofen — Intravenous ibuprofen will be administered for treatment of pain in adults presenting to the ED with biliary colic
  Other Names: Caldolor; NeoProfen
  Arms: IV Ibuprofen: Adults age 18-55 years
Drug: Saline — Saline will be administered to the placebo group
  Arms: Control Group: Adults age 18-55 years

SUMMARY:
The aim of this study is to assess the analgesic efficacy of intravenous ibuprofen given in the Emergency Department for the treatment of biliary colic. We hypothesize that intravenous ibuprofen will provide a clinically significant drop in self-reported patient pain level as measured by the visual analog scale.

DETAILED DESCRIPTION:
It is estimated over 20 million people aged 20-74 have gallbladder disease, with biliary colic being a common and painful symptom in these patients. Likely due to the relatively recent approval of intravenous ibuprofen use for fever and pain in adults, no assessment of its analgesic efficacy for biliary colic currently exists in the literature.

Utilizing a visual analog scale (VAS) for patient self-assessment of pain, this study will address this lack of evidence and identify intravenous ibuprofen's value as a novel analgesic in the treatment of biliary colic. Patients will be given a VAS at the time of study therapy administration, at 15-minute intervals during the first hour post-administration, and 30-minute intervals in the second hour. Though NSAID's have been extensively studied in the management of this phenomenon, this study aims to help optimize pain treatment of patients presenting to the Emergency Department with biliary colic, and potentially pave the way for future analgesic treatment comparison studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18-55
* Present to ED with right upper quadrant (RUQ) abdominal pain
* Suspected diagnosis of biliary colic
* Negative pregnancy test for women of childbearing potential (complete POC testing form)
* No history of cholecystectomy

Exclusion Criteria:

* Patient age < 18 or > 55
* Incarcerated
* Hemodynamic instability
* Inability to reliably self-report or communicate pain intensity and pain relief
* Taking Warfarin
* Cannot consent of are not competent to consent
* Hepatic, renal, cardiac failure
* NSAID or morphine allergy
* History congenital bleeding diathesis or platelet dysfunction
* Peptic ulcer diseases
* Are otherwise unsuitable for the study in the opinion of the investigator/sub-investigators

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-09-09 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Quan, DO, Principal Investigator — Valleywise Health
Locations (1):
- Maricopa Integrated Health System, Phoenix, Arizona, United States

REFERENCES:
- [Background] Promes JT, Safcsak K, Pavliv L, Voss B, Rock A. A prospective, multicenter, randomized, double-blind trial of IV ibuprofen for treatment of fever and pain in burn patients. J Burn Care Res. 2011 Jan-Feb;32(1):79-90. doi: 10.1097/BCR.0b013e3182037300. PMID 21127424
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Krudsood S, Tangpukdee N, Wilairatana P, Pothipak N, Duangdee C, Warrell DA, Looareesuwan S. Intravenous ibuprofen (IV-ibuprofen) controls fever effectively in adults with acute uncomplicated Plasmodium falciparum malaria but prolongs parasitemia. Am J Trop Med Hyg. 2010 Jul;83(1):51-5. doi: 10.4269/ajtmh.2010.09-0621. PMID 20595477
- [Background] Morris PE, Promes JT, Guntupalli KK, Wright PE, Arons MM. A multi-center, randomized, double-blind, parallel, placebo-controlled trial to evaluate the efficacy, safety, and pharmacokinetics of intravenous ibuprofen for the treatment of fever in critically ill and non-critically ill adults. Crit Care. 2010;14(3):R125. doi: 10.1186/cc9089. Epub 2010 Jun 30. PMID 20591173
- [Background] Singla N, Rock A, Pavliv L. A multi-center, randomized, double-blind placebo-controlled trial of intravenous-ibuprofen (IV-ibuprofen) for treatment of pain in post-operative orthopedic adult patients. Pain Med. 2010 Aug;11(8):1284-93. doi: 10.1111/j.1526-4637.2010.00896.x. Epub 2010 Jun 30. PMID 20609131
- [Background] Kroll PB, Meadows L, Rock A, Pavliv L. A multicenter, randomized, double-blind, placebo-controlled trial of intravenous ibuprofen (i.v.-ibuprofen) in the management of postoperative pain following abdominal hysterectomy. Pain Pract. 2011 Jan-Feb;11(1):23-32. doi: 10.1111/j.1533-2500.2010.00402.x. PMID 20642488
- [Background] Southworth S, Peters J, Rock A, Pavliv L. A multicenter, randomized, double-blind, placebo-controlled trial of intravenous ibuprofen 400 and 800 mg every 6 hours in the management of postoperative pain. Clin Ther. 2009 Sep;31(9):1922-35. doi: 10.1016/j.clinthera.2009.08.026. PMID 19843482
- [Background] Smith HS, Voss B. Pharmacokinetics of intravenous ibuprofen: implications of time of infusion in the treatment of pain and fever. Drugs. 2012 Feb 12;72(3):327-37. doi: 10.2165/11599230-000000000-00000. PMID 22316349
- [Background] Colli A, Conte D, Valle SD, Sciola V, Fraquelli M. Meta-analysis: nonsteroidal anti-inflammatory drugs in biliary colic. Aliment Pharmacol Ther. 2012 Jun;35(12):1370-8. doi: 10.1111/j.1365-2036.2012.05115.x. Epub 2012 Apr 29. PMID 22540869
- [Background] Henderson SO, Swadron S, Newton E. Comparison of intravenous ketorolac and meperidine in the treatment of biliary colic. J Emerg Med. 2002 Oct;23(3):237-41. doi: 10.1016/s0736-4679(02)00524-3. PMID 12426013
- [Background] Olsen JC, McGrath NA, Schwarz DG, Cutcliffe BJ, Stern JL. A double-blind randomized clinical trial evaluating the analgesic efficacy of ketorolac versus butorphanol for patients with suspected biliary colic in the emergency department. Acad Emerg Med. 2008 Aug;15(8):718-22. doi: 10.1111/j.1553-2712.2008.00178.x. Epub 2008 Jul 11. PMID 18637080

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Saline-only control group
  Saline: Saline will be administered to the placebo group
- IV Ibuprofen: Patients receiving intravenous ibuprofen therapy
  IV Ibuprofen: Intravenous ibuprofen will be administered for treatment of pain in adults presenting to the ED with biliary colic
Period: Overall Study
Arm/Group | Control Group | IV Ibuprofen
Started | 11 | 11
Completed | 9 | 9
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline data for the population is VAS pain score prior to Intravenous Ibuprofen or Placebo administration.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | IV Ibuprofen | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Customized [Count of Participants; unit: Participants] — Ages 18-55 were enrolled. Individual subject's age data was not reported. Population: Age for subjects analyzed.
  Participants
    18-55 years of age: number analyzed (Participants) | 9 | 9 | 18
    18-55 years of age | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Male or Female for participants analyzed.
  Participants
    Female | 8 | 7 | 15
    Male | 3 | 4 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Pain score [Mean (Standard Deviation); unit: units on a scale] — Visual Analog pain score where 0=no pain, and 10=worse pain imaginable.
  units on a scale | 5 (0.015) | 6 (0.029) | 6 (0.001)

OUTCOME MEASURES:

1. Primary Outcome: Pain Score 120 Minutes After Study Medication Administration
Description: Pain is measured on a visual analog scale 0=no pain and 10=worst pain imaginable.
Time Frame: 120 minutes post medication administration
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control Group: Adults Age 18-55 Years | IV Ibuprofen: Adults Age 18-55 Years
Number analyzed (Participants) | 9 | 9
score on a scale | 3.0 [0.0 to 7.0] | 0.3 [0.0 to 8.0]

ADVERSE EVENTS:
Time Frame: During study treatment (about 2 hours).
Arm/Group | Control Group | IV Ibuprofen
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
There were not enough patients enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT02268955/Prot_SAP_000.pdf